CLINICAL TRIAL: NCT05645068
Title: Pilot Study for the Evaluation of Retinal Microvasculature by OCT Angiography During a Multidisciplinary Management Program Integrating Physical Activity in Type 2 Diabetic Subjects.
Brief Title: Retinal Microvasculature by Optical Coherence Tomography Angiography During Integrating Physical Activity in Diabetic Subjects.
Acronym: OCTACTIPH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/21/0612; 2022-A02003-40 (Other: ID-RCB)
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Complications
Keywords: Optical Coherence Tomography Angiography; Diabetic Macular Edema
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optical Coherence Tomography Angiography (Experimental)
  Interventions: Diagnostic Test: Optical Coherence Tomography Angiography; Other: multidisciplinary care program

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography Angiography — Optical Coherence Tomography Angiography
Other: multidisciplinary care program — multidisciplinary care program including sports activity

SUMMARY:
Diabetic retinopathy is a common condition of diabetes and can lead to blindness, making it one of the most feared complications of diabetes.

Recently, it has been proven that the parameters measured by Optical Coherence Tomography (OCT) Angiography: the vascular density of the macular retinal capillary plexi and the foveolar avascular zone, can be modified after a high-intensity sports training program in healthy subjects.

the team wants to study the evolution of the macular, in type 2 diabetic subjects, before and after a stay in a care structure dedicated to the multidisciplinary and integrative management (nutrition, physical activity, therapeutic education) of a duration of 3 weeks.

DETAILED DESCRIPTION:
The prevention of vascular and neurological complications in diabetic subjects represents a major public health issue. Diabetic retinopathy is a common condition of diabetes and can lead to blindness, making it one of the most feared complications of diabetes.

Diabetes management is global and aims at a stable glycemic balance putting the patient out of the micro and macrovascular complications linked to this pathology. It involves modifying the lifestyle of patients with the practice of appropriate physical activity, balancing daily food intake, not necessarily by taking insulin-sensitizing or hypoglycemic drug treatment, but also by management of other risk factors related to complications: dyslipidemia, weight, smoking, arterial blood pressure balance.

The use of Optical Coherence Tomography Angiography allow the evaluation of the microvasculature of the macula.

Diabetic macular edema is the leading cause of vision loss in type 2 diabetic subjects mainly due to dysfunction of the macular microvasculature.

Macular analysis via Optical Coherence Tomography Angiography can quickly and non-invasively predict the risk of occurrence of Diabetic macular edema and therefore that of a decrease in acuity and visual impairment.

ELIGIBILITY:
Inclusion Criteria:

* Patient for whom a 3-week multidisciplinary and integrative program was offered in a diabetology unit
* Patient having given his consent
* Patient affiliated to a social security scheme or equivalent
* Patient with type 2 diabetes

Exclusion Criteria:

* History of exudative or tractional retinal detachment
* Intraocular foreign body
* History of endophthalmitis
* History of inflammatory disease of the retina
* History of chorioretinitis
* Patient with age-related macular degeneration
* Patients with type 1 diabetes or secondary diabetes
* Uncontrolled hypertension does not define Systolic arterial pressure (SAP) > 180 mmHg or Diastolic arterial pressure (DAP) > 110 mmHg
* Patient who has already received intravitreal injections of anti-angiogenic molecules.
* Pregnant or breastfeeding patient at the time of the study
* Persons under a legal protection regime for adults (safeguard of justice, guardianship, curatorship, institutionalized, or under mandate for future protection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
coefficient of variation of the superficial retinal capillary plexus | week 3
  coefficient of variation of the superficial retinal capillary plexus between day 0 and week 3 determinate by OCT Angiography

CONTACTS AND LOCATIONS:
Overall Officials: Fanny VARENNE, PH, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No